### **Diabetes Prevention Program Feasibility Study of Breastfeeding**

Principal Investigator: Lisette Jacobson, PhD, MPA, MA

Mentors: Tracie Collins, MD, MPH, MHCDS; David Robbins, MD; Judy Stern, PhD

Key Personnel: David Grainger, MD, MPH; Kelsey Lu, MS; Meredith Lucas, BA; Hayrettin Okut, PhD; Niaman Nazir, MBBS, MPH; Michael Wolfe, MD; Rosey Zackula MA

Consultants: Brenda Bandy, IBCLC; Jolynn Dowling, MSN, APRN, NNP-BC, IBCLC

Version: March 25, 2019

### Section I. Purpose, Background and Rationale

### A. Specific Aims and Hypotheses

In the proposed randomized controlled trial, we seek to determine the feasibility and efficacy of a combined breastfeeding, DPP-based program in a cohort of overweight/obese women to be followed during pregnancy through 6 months postpartum. Our trial will have three study arms: DPP plus breastfeeding (Tx1); DPP Only (Tx2); and Usual Care (Tx3). Specific aims are:

<u>Aim 1</u>: Test the efficacy of Tx1 to improve 6-month postpartum weight loss among women with a BMI  $\geq$  25. We will measure maternal height and weight at baseline; weight at delivery and 6 months postpartum.

<u>Hypothesis 1</u>: Women in Tx1 will have greater weight loss postpartum compared to women in Tx2 and Tx3.

<u>Aim 2</u>: Test the efficacy of Tx1 to improve 6-month postpartum mean blood glucose (HbA1c) and mean arterial blood pressure among women with a BMI  $\geq$  25. We will measure HbA1c and mean arterial blood pressure at baseline, delivery, and 6 months postpartum. <u>Hypothesis 2</u>: Women in Tx1 will have better HbA1c and mean arterial blood pressure postpartum compared to women in Tx2 and Tx3.

Aim 3: Test the efficacy of Tx1 to increase any breastfeeding through 6 months postpartum among women with a BMI  $\geq$  25. We will measure any breastfeeding continuance at week 1, 3, and 6 postpartum, and at 3 and 6 months.

Hypothesis 3: Women in Tx1 will breastfeed longer compared to women in Tx2 and Tx3.

# B. Background and Significance

Gestational diabetes mellitus (GDM) affects between 6%<sup>1-3</sup> to 20%<sup>2,4</sup> of pregnant women in the United States. Overweight and obesity are a major risk factor for GDM<sup>5-9</sup> and also considered an independent risk factor for other adverse health outcomes.<sup>10-15</sup> Women with a history of GDM have at least a seven-fold increased risk of developing type 2 diabetes mellitus (T2DM) compared to women who do not have GDM.<sup>16,17</sup> Gestational diabetes is associated with increased maternal and neonatal morbidity and mortality.<sup>18-29</sup> Complications of GDM are further increased for rural women who often experience limited access to obstetrical healthcare services,<sup>30-33</sup> leading to poor birth outcomes<sup>34-36</sup> and reduced breastfeeding rates.<sup>37</sup>

Against this background, we completed a pilot health assessment in a rural southwest Kansas community with an alarming number of high-risk pregnancies complicated by gestational diabetes, 11% vs. 6% nationally.<sup>2</sup> Half of respondents were Hispanic of low socio-economic status.<sup>38</sup> During pregnancy, three-quarters of women were overweight/obese, did not exercise, and had a family history of diabetes.<sup>38</sup> Further, findings from a qualitative follow-up study within this same community indicated that women had limited access to health promotion programs and breastfeeding services.

Rural communities with limited availability of health promotion programs and potentially high rates of chronic disease face a myriad of problems. First, diabetes is associated with adverse health outcomes for mother and child. Women with GDM are at increased risk for pregnancy and delivery complications — including preeclampsia, 18-22 cesarean section, 18,19,22,23 pregnancyinduced hypertension, <sup>20,23,28</sup> preterm birth, <sup>19,20</sup> shoulder dystocia, <sup>18,20,24</sup> and macrosomia <sup>18,20,22</sup>-27,29 — leading to increased maternal and neonatal morbidity and mortality. 18,24,29,39 Infants born to mothers with GDM are more likely to have neonatal hypoglycemia, <sup>26,40</sup> hyperinsulinemia, <sup>26,40</sup> and are at greater risk for developing metabolic syndrome, 41 diabetes, 42 and obesity during childhood/adolescence. 43-45 Second, having a pregnancy complicated with GDM and residing in a rural location is particularly challenging due to limited access and availability of healthcare services. 46-51 Specifically, rural pregnant women have a higher likelihood of low birth-weight babies and pre-term delivery, <sup>30,34-36</sup> high smoking rates, <sup>37,52</sup> and reduced breastfeeding rates. <sup>37</sup> Due to geographic barriers, high rates of chronic disease including obesity, and limited availability of health promotion programs coupled with a demonstrated need for health behavior change, it becomes important to test an intervention during the prenatal and postnatal period among this at-risk population. This period is particularly conducive to behavior change because: (1) women are more likely to modify their behavior to benefit their children, (2) behavior change interventions are most successful in the short term, and (3) effective interventions that start during pregnancy are more likely to be sustained after birth, thereby reducing the risk of retaining excess weight and maternal obesity. 53,54

Given the demonstrated need for health behavior change, it is worthwhile to test the use of an intervention during the prenatal and postnatal period. The Diabetes Prevention Program (DPP) is associated with a reduced risk of developing T2DM by 58% through counseling on effective

diet, exercise, and behavior modification.<sup>55</sup> There is also evidence to support the use of this efficacious program in reducing postpartum weight.<sup>56,57</sup> Further, recent evidence suggests that longer duration of breastfeeding is associated with lowering T2DM incidence,<sup>58-61</sup> reducing maternal postpartum weight,<sup>62-64</sup> and resetting maternal metabolism after pregnancy.<sup>65</sup> Breastfeeding also protects against breast cancer,<sup>66</sup> ovarian cancer,<sup>67,68</sup> and T2DM.<sup>69,70</sup> Despite these findings, no studies have addressed the role of intensive breastfeeding support combined with an efficacious weight loss program to reduce postpartum weight, thereby reducing progression to T2DM after pregnancy.

The American Academy of Pediatrics<sup>71</sup> and the World Health Organization<sup>72</sup> recommend breastfeeding for the first 6 months of life. In Kansas,  $79\%^{73}$  of women with a BMI  $\geq 25$  start breastfeeding, and only  $29\%^{73}$  still breastfeed with some supplementation (defined as "any breastfeeding") at 6 months postpartum. The Kansas rate for high BMI women of 29% is unacceptable and an urgent public health concern when compared to the 6-month breastfeeding rate for normal BMI Kansas women of 51% and the Healthy People 2020 goal of 61%.<sup>74</sup> In the proposed randomized controlled trial, we seek to determine the feasibility and efficacy of a combined breastfeeding, DPP-based program in a cohort of overweight/obese women to be followed during pregnancy through 6 months postpartum. Our trial will have three study arms: DPP plus breastfeeding (Tx1); DPP Only (Tx2); and Usual Care (Tx3). A total sample of 60 pregnant women in their 1st or 2nd trimester with a BMI  $\geq 25$  will be recruited. Eligible participants are randomly assigned to a study arm (20 per arm).

### C. Preliminary Studies

I led and completed two pilot studies in southwest rural Kansas: (1) a health assessment of the obstetrical population (completed in April 2015), and (2) a follow-up focus group study with the same population (completed in May 2016). The purpose of the assessment was to learn about the health behaviors of rural pregnant women. Two local hospitals and one federally qualified rural health center participated in the assessment. Our sample consisted of 177 rural pregnant women. Key findings indicated that the majority of women were Hispanic (50.3%), 18-25 years old (48.6%), high school educated (51.2%), WIC enrolled (51.7%), and earned < \$25,000/year (54.2%).<sup>38</sup> The majority were overweight (28.1%) or obese (26.2%) *prior* to pregnancy, which increased to 34.4% and 41.6% respectively during pregnancy.<sup>38</sup> Additionally, the majority engaged in no daily exercise (72.6%) and nearly one-third (30.5%) reported having an immediate family member who was diagnosed or treated for diabetes or cardiovascular disease.<sup>38</sup> These results demonstrate significant diabetes risk factors during and after pregnancy. Subsequently, in follow-up to the assessment, I led and completed a focus group study to gain in-depth information from this same population on what they would value in a health promotion program. Findings indicated limited availability of programs that focus on exercise, diet, and breastfeeding support during and after pregnancy. Further, I published three additional studies relevant to the proposed project.<sup>37,52,75</sup> Each of these studies focused on health behaviors among urban versus rural WIC enrolled women in Kansas and helped our research team understand the prenatal and postnatal needs of at-risk populations in Kansas. These studies also provided me with

experience in collaborating with other researchers and with the process of publishing a manuscript in a high-impact professional journal.

### D. Rationale for Proposed Study

Risk factors for diabetes are well documented.<sup>5-9</sup> Maternal obesity in particular increases the risk of negative health outcomes for mother<sup>15,76-80</sup> and child, <sup>81-86</sup> including the propensity for women to retain excessive postpartum weight leading to obesity in subsequent pregnancies. 87-90 Less is known about protective factors relevant to diabetes though evidence suggests that longer duration of breastfeeding among women with a history of GDM is associated with lower incidence of developing type 2 diabetes up to two years after pregnancy. 58-61 Breastfeeding also appears to lower maternal postpartum weight<sup>62-64</sup> and facilitates the resetting of maternal metabolism after pregnancy. 65 The Diabetes Prevention Program (DPP) is associated with a reduced risk of developing diabetes by 58%<sup>55</sup> and there is evidence to support the use of this efficacious program in reducing postpartum weight. <sup>56,57</sup> Despite these findings, no studies have used a DPP-enhanced version that includes intensive breastfeeding counseling and support for overweight and obese women. Given that overweight and obese women at risk for GDM are also less likely to start and continue breastfeeding, 84,91-93 it is critical that interventions for reducing GDM risk also include breastfeeding support that is uniquely tailored to the needs of this population. This is where the current proposal narrows the gap and contributes to the body of knowledge about reducing diabetes risk factors during and after pregnancy in an underserved population with scarce healthcare resources available.

# E. Impact of Proposed Study

The proposed project will inform future intervention efforts that aim to reduce diabetes risk factors during and after pregnancy and to increase breastfeeding, thereby improving short- and long-term maternal and child health outcomes. The <u>immediate impact</u> will be to reduce diabetes risk factors among a high-risk population and inform interventions aimed at reducing these risk factors and decreasing disproportionate morbidity. Its <u>ultimate potentially high public health impact</u> is GDM and type 2 diabetes prevention among a racially and ethnically diverse, at-risk population.

### F. Justification for Project

Risk factors for diabetes are well documented,<sup>5-9</sup> but less is known about some factors that attenuate the risk for GDM. Recent studies support the use of the Diabetes Prevention Program in reducing postpartum weight.<sup>56,57</sup> Moreover, emerging research suggests that longer duration of breastfeeding among women with a history of GDM decreases the likelihood of developing type 2 diabetes within two years after pregnancy.<sup>58-61</sup> However, no prior studies have assessed the feasibility and efficacy of a DPP-based intervention that includes intensive breastfeeding counseling and support among racially and ethnically diverse reproductive-age rural women. Rural pregnant women in particular have decreased access to healthy foods and fewer options to engage in physical activity.<sup>94-98</sup> Furthermore, Hispanic women often supplement breastfeeding with formula, triggering decreased milk supply and early breastfeeding cessation.<sup>99-101</sup> The

proposed research is *innovative* because it represents a departure from what has been accomplished in the field thus far: *We seek to implement a combined breastfeeding, DPP-based intervention and determine its feasibility and efficacy as well as its effect on metabolic outcomes among an at-risk population. Through examination of postpartum weight, breastfeeding behavior, and metabolic markers, results of the proposed project will inform the development of interventions to reduce diabetes risk factors during and after pregnancy. Furthermore, an efficacious approach toward promoting exercise, nutrition, and breastfeeding can be integrated into the continuum of healthcare services provided to racially and ethnically diverse, at-risk rural pregnant women.* 

## Section II. Research Plan and Design

#### A. Study Design Overview Figure 1. Study Design Screen individuals for eligibility After meeting study inclusion criteria, randomize individuals into Tx1, Tx2, or Tx3 Tx2 Tx3 Intervention (Tx1) **DPP** plus **DPP Only Usual Care** Breastfeeding (N=20) (N=20) (N=20) Ρ DPP - 16 sessions: Core Regular prenatal care DPP - 16 sessions: R R provided by physician curriculum (Phase I) Core curriculum (Phase I) E Е **Breastfeeding Education** N Ν 2-hour curriculum Α Α (between weeks 20 - 24) т т Breastfeeding Booster Α Α Session 1-hour curriculum L L (between weeks 28 - 32) Р At delivery – in-hospital At delivery - in-hospital At delivery - in-hospital 0 breastfeeding support breastfeeding support breastfeeding support s DPP - 15 sessions: Post-DPP - 15 sessions: Т core curriculum (Phase II) Post-core curriculum N (Phase II) Α **Breastfeeding** т Т Assessment (at five Α Α separate time points)

This is a three-arm pilot randomized controlled trial (RCT) to implement as well as determine the feasibility and efficacy of an intervention that is based on the Diabetes Prevention Program and includes intensive breastfeeding counseling and support among a cohort of overweight and obese pregnant women. Upon meeting eligibility criteria, participants will be randomly assigned to the DPP plus breastfeeding (intervention, Tx1), DPP Only (Tx2), or Usual Care (Tx3), and will be followed during pregnancy through 6 months postpartum. Participants in Tx1 will receive the DPP and targeted breastfeeding support during pregnancy through 6 months postpartum. Participants in Tx2 will receive the DPP only. Participants in

Tx3 will receive care as usual. Usual care is described as obstetrical care that women with normal BMI receive and that is provided by the same provider (Dr. Michael Wolfe).

At recruitment and at study closure, participants will complete four survey instruments; each of which assesses women's knowledge of physical activity, nutrition, and breastfeeding (see appendices 1 through 4). Also, postpartum women will complete the Edinburgh Postnatal Depression Scale (EPDS, see appendix 5) and a study coordinator will assess postpartum women's breastfeeding experience with the Bristol Breastfeeding Assessment Tool (BBAT, see

appendix 6). Weight, mean blood glucose (HbA1c), mean arterial blood pressure, and glucose tolerance levels during pregnancy as well as initiation and duration of breastfeeding will be measured for all participants through 6 months postpartum.

### **B.** Duration of Study

It is anticipated that after receiving Institutional Review Board (IRB) approval, recruitment will begin during the last quarter of 2019 and will continue through June of 2020. We will recruit over a period of 9 months and the last follow up with women will take place at 6 months postpartum. The trial will be completed over a 24-month period and will conclude during the second quarter of 2021. Data collection and preliminary data analysis will take place as the trial runs. Final data analysis and dissemination of findings will all take place following completion of the trial, during 2021 and 2022.

### C. Number of Participants

This IRB protocol pertains to the recruitment of eligible participants from two obstetrical clinics: one clinic at Via Christi Health (VCH), a regional hospital in Wichita, and another clinic at Kearny County Hospital, a full-service hospital in rural southwest Kansas. About 45% (16,797) of Wichita's Hispanic population is female and of reproductive age, 102 and the VCH clinic sees a high volume of this at-risk population at an average of 123 pregnant patients per month, with an average pre-pregnancy BMI of 30.5 (personal communication by senior management staff at VCH on January 18, 2017). These socio-demographic and health data are similar to those of atrisk rural pregnant women in southwest Kansas who visit Kearny County Hospital (KCH) for prenatal and postnatal care. Dr. Michael Wolfe, maternal fetal medicine specialist, sees pregnant women at both of these locations (VCH and KCH), and he and his staff will actively assist with patient recruitment. Our goal is to randomize a total of 72 eligible participants (24 women in each study arm, which translates to 12 women from each recruitment site). Our recruitment target of overweight or obese pregnant women will involve 50% Hispanic women (who are English-speaking) and 50% other race including non-Hispanic whites. The population of pregnant women in southwest Kansas who deliver at Kearny County Hospital, Lakin, Kansas, is estimated to be 300 individuals, of which 75% (or 225 individuals) have a BMI  $\geq$  25 and  $\leq$  35.

### D. Subject Selection Criteria and Recruitment

We will recruit pregnant patients from two obstetrical clinics: one clinic at Via Christi Hospitals Wichita, Inc. (VCH), a regional hospital in Wichita, and another clinic at Kearny County Hospital, a full-service rural hospital located in Lakin, southwest Kansas. Dr. Michael Wolfe, maternal fetal medicine specialist, sees pregnant women at this location, and he and his staff will actively assist with patient recruitment. During the first prenatal appointment, Dr. Wolfe will screen potential participants for inclusion criteria, and if he believes a participant meets inclusion criteria (see Table 1), then he will familiarize a potential participant with the study's purpose. If the potential participant is interested in the study, then he will give her a study brochure and a hard copy of the consent form. Prior to using this study brochure, the brochure will be reviewed and approved by the IRB at Via Christi Hospitals Wichita, Inc. By providing the potential

participant with a copy of the consent form, this will serve as the verbal consent script. Dr. Wolfe will also provide the potential participant's name and phone number to Dr. Jacobson and her research coordinator. After receiving a potential participant's name and phone number from Dr. Wolfe, the research coordinator will follow up with a phone call to determine if the potential participant again meets study inclusion criteria, and if she does, the coordinator will screen if the potential participant meets study exclusion criteria during the same phone call (see Table 1). Before the research coordinator screens for inclusion and exclusion criteria, during this same phone call, verbal consent will be obtained between the participant and the research coordinator, using the consent form as the verbal consent script, and then written e-consent will be obtained via REDCap at the orientation session. Once the participant is enrolled in the study and over the course of her pregnancy develops one of the conditions mentioned under Exclusion (Table 1), then this will be reported to the Data and Safety Officer. It will then be decided in consultation with Dr. Wolfe if the participant will be able to continue participating in the study or if she will need to be dismissed.

Table 1. Enrollment Criteria

| <del></del> |
|----------------------------------------------------------|
| Inclusion |
| 1. Pregnant |
| 2. In 1st trimester or early in 2nd trimester |
| 2. BMI ≥ 25 and < 35 |
| 3. At least 18 years old or older |
| Be able to understand English |
| 5. Must have a cell phone |
| 6. Able to use Facebook |
| 7. Able to use Skype, FaceTime or Zoom |
| Exclusion |
| Pregnancy complications that require emergency care |
| 2. Thyroid disease |
| 3. Multiple gestation |
| 4. Substance abuse within last 3 years |
| 5. ART (Assisted Reproductive Technology) pregnancy |
| 6. Current smoker |
| 7. Prior bariatric surgery |
| 8. In weight-loss program within 3 months of conception |
| 9. BMI ≥ 35 |
| 10. Unable to attend intervention/follow-up visits |
| 11. Unwilling to self-monitor data collection |
| 12. Unable to complete intervention |
| 13. Presence of any condition that limits walking |
| 14. Presence of any condition that limits following diet |
| recommendations |
| 15. Pregnancies complicated with fetuses diagnosed with |
| lethal malformations/conditions |

If the participant meets enrollment criteria, then the research coordinator will call her again to assign her a time and place for the orientation session, to complete study-related survey instruments, and to obtain her email address to provide her with informed consent materials for review. Participants are informed that they will earn incentives to continue and complete the study: (1) a \$50 gift card at study entry, (2) a digital scale and pedometer at delivery, and (3) a gift up to \$75 for baby at Walmart's baby registry at study closure. Investigators will issue incentives in accordance with policies set forth by

IRB (please refer to the heading titled "Self-Administered Surveys and Incentive to Participate" below for additional detail regarding participant incentives).

Our recruitment target of overweight or obese pregnant women will involve 50% Hispanic women (who are English-speaking) and 50% other race including non-Hispanic whites. We anticipate meeting our recruitment goals through multiple approaches. We will promote the study via targeted mailings and clinic posters. We will advertise and develop study materials in English only. We will recruit over a period of 9 months, planning to randomize 2-3 participants

each week, or 1-2 participants per site. Our goal is to randomize a total of 72 pregnant women (24 women in each study arm, 12 women per site). Given an attrition rate of 20%, this will leave us with 60 women total (20 women in each study arm, or 10 women per site in each study arm).

### **E. Study Locations**

Recruitment will take place at two obstetrical clinics: 1) Via Christi Hospitals Wichita, Inc., Kansas, and 2) Kearny County Hospital, Lakin, Kansas. We will have on-going support from both hospitals. Michael Mullins, Senior Vice President, Ascension Healthcare and Laurie Labarca, Hospital President St. Joseph, Via Christi Hospitals Wichita, Inc. as well as Benjamin Anderson, Chief Executive Officer Kearny County Hospital, fully support Dr. Jacobson's work to determine the feasibility and efficacy of a combined breastfeeding, DPP-based program in a cohort of overweight/obese women to be followed during pregnancy through 6 months postpartum (see their letters of support, Appendix 7-8). Most importantly, we will have ongoing support for Dr. Jacobson's work from Dr. Michael Wolfe, Maternal Fetal Medicine Specialist, who sees pregnant women at both locations (see letter of support, Appendix 9).

Locations for each obstetrical clinic affiliated with the hospitals above are as follows:

Kearny County Hospital

500 East Thorpe Street

Lakin, Kansas 67860

Via Christi Maternal Fetal Medicine Clinic
1515 South Clifton Avenue, Suite 130
Wichita, Kansas 67218

# F & G. Methodology - Intervention, Study Procedures and Data Collection

#### **The Intervention**

Conceptual Model. We will use Social Cognitive Theory (SCT)<sup>103,104</sup> and Self-Determination Theory (SDT)<sup>105,106</sup> to guide program development and selection of measures. SCT stipulates that behavior modification results from the interaction between behavior change, cognition (self-efficacy, perception of barriers to lifestyle changes), and the environment (support), while modeling and reinforcement serve to encourage change. SDT is a broad-based theory of human motivation<sup>107</sup> that explains how intrinsic motivation can lead to improve eating and exercise patterns.<sup>108</sup> According to SDT, a person's increased intrinsic motivation to improve eating and exercise patterns should positively relate to self-efficacy and the ability to overcome barriers and solicit support. The DPP plus breastfeeding (Tx1) uses assignments, individualized goal setting, and shared problem-solving to increase mastery and goal achievement in incremental steps to enhance self-regulatory skills.

**Diabetes Prevention Program (DPP).** Dr. Jacobson and the research coordinator will administer the DPP in two phases. <u>Phase I</u> consists of a total of 16 sessions that will be completed during pregnancy (see Table 2). Two of the Phase I DPP sessions have been replaced with the <u>Cooking Matters</u><sup>47</sup> curriculum: DPP session #2 has been replaced with creating a healthy home food environment, and DPP session #4 with incorporating more fruits, vegetables,

and whole grains into family meals. <u>Cooking Matters</u> empowers low-income families with the skills to cook healthy, affordable meals at home. Its curriculum uses the Dietary Guidelines for Americans<sup>109</sup> and MyPlate<sup>71</sup> as the foundation for basic nutrition guidelines. Each of the sixteen (16) sessions/modules of Phase I will be pre-recorded and archived on a secure, private group on Facebook. Only Tx1 and Tx2 participants, Dr. Jacobson and the research coordinator will have access to this Facebook group.

We will employ a "rolling" recruitment period of 9 months, meaning that each participant may be at different completion stages. During their first face-to-face orientation session, participants will receive access to the secure, private group on Facebook. They will be asked to complete each Phase I module on their own time, starting at week 19 of pregnancy. To supplement their self-study of the curriculum, on a weekly basis, the research coordinator will follow up with each study participant via phone to check on progress. If participants do not make adequate progress, then the coordinator will assess how much extra time the participant needs to complete a module, and will work with her face-to-face via Skype, FaceTime or Zoom if needed. Participants will complete Phase I by week 33 of pregnancy.

<u>Phase II</u> consists of a total of 15 sessions that will be completed after delivery (see Table 2). Two of the Phase II DPP sessions (sessions #4 and #5 respectively) have been modified with the <u>Cooking Matters</u> curriculum that (1) emphasizes planning/preparing for healthy, low-cost meals and (2) encourages mothers to make smart choices when food shopping. Each of the fifteen (15) sessions/modules of Phase II will be pre-recorded and archived on the same secure, private group on Facebook mentioned above. Only Tx1 and Tx2 participants, Dr. Jacobson and the research coordinator will have access to this Facebook group.

Participants will re-engage into the DPP with another face-to-face orientation session conducted by Dr. Jacobson at week 6 postpartum. The same session completion format and procedure for inadequate progress will be followed as during pregnancy. Participants will complete <a href="Phase II">Phase II</a> by week 20 postpartum. An 80% completion rate of each phase is considered successful completion of the intervention.

Table 2. Timetable - Diabetes Prevention Program Sessions

| Prenatal (Core Curriculum) | Postnatal (Post-core Curriculum) | | |
|---|---|---|---|
| | Week of | | Week of |
| DPP Sessions - Phase I | Pregnancy | DPP Sessions - Phase II | Postpartum |
| 1 - Orientation - Welcome! | 18 | 1 - Orientation - Welcome Back! | 6 |
| 2 - Cooking Matters (CM): Set a Healthy Example | 19 | 2 - Fats: Saturated, Unsaturated, & Trans-Fats | 7 |
| 3 - Eating Less Fat and Fewer Calories | 20 | 3 - Food Preparation & Recipe Modification | 8 |
| 4 - CM: Choosing Fruits, Vege's, Whole Grains | 21 | 4 - Taking It One Meal at a Time, CM: Planning | 9 |
| 5 - Move Those Muscles | 22 | 5 - Variety and Balance, CM: Shopping | 10 |
| 6 - Being Active - A Way of Life | 23 | 6 - More Volume, Fewer Calories | 11 |
| 7 - Tip the Calorie Balance | 24 | 7 - Staying on Top of Physical Activity | 12 |
| 8 - Take Charge of What's Around You | 25 | 8 - Stepping Up to Physical Activity | 13 |
| 9 - Problem Solving | 26 | 9 - Long-term Maintenance | 14 |
| 10 - Four Keys to Healthy Eating Out | 27 | 10 - Holidays, Vacations, Special Events | 15 |
| 11 - Talk Back to Negative Thoughts | 28 | 11 - Preventing Relapse | 16 |
| 12 - The Slippery Slope of Lifestyle Change | 29 | 12 - Stress and Time Management | 17 |
| 13 - Jump Start Your Activity Plan | 30 | 13 - Heart Health | 18 |
| 14 - Make Social Cues Work for You | 31 | 14 - A Closer Look at Type 2 Diabetes | 19 |
| 15 - You Can Manage Stress | 32 | 15 - Looking Back and Looking Forward | 20 |
| 16 - Ways to Stay Motivated | 33 | | |

**Breastfeeding.** Additionally, participants in Tx1 will receive an educational session on breastfeeding and will register for and participate in a professional peer support group (see Table 3). Participants in Tx2 and Tx3 will not receive breastfeeding education or register/participate in a professional peer support group. The 2-hour breastfeeding session is pre-recorded into four (4) 30-minute sessions and archived on the same secure, private Facebook group as mentioned previously. Participants will have access to all four breastfeeding sessions by week 24 of pregnancy and they need to complete all sessions by week 30 of pregnancy. The breastfeeding session will be taught by an International Board Certified Lactation Consultant (IBCLC).

At delivery, all participants will receive some type of lactation support in the hospital. However, only participants in Tx1 will be provided with a breastfeeding assessment at day 3, day 10, week 3 and week 6, as well as months 2, 3 and 6 postpartum (see Table 3). The breastfeeding telephone assessment is modelled after the Bristol Breastfeeding Assessment Tool (BBAT)<sup>110</sup> (see Appendix 6) and used to improve an infant's positioning, attachment, sucking, and swallowing. During these telephone assessments, Dr. Jacobson's research coordinator will assess if mother and baby need breastfeeding support from a lactation professional. If the telephone assessment warrants an in-person visit, then the research coordinator will put mother and baby in contact with a lactation professional provided by the hospital.

Table 3. Breastfeeding Support for Women in Tx1 (Intervention Arm) Only

| | Prenatal | Postnatal | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Intervention Components | Week 24 - 30 | Day 3 | Day 10 | 3 Weeks | 6 Weeks | 2 Months | 3 Months | 6 Months |
| Breastfeeding Education (2-hour curriculum) | X | | | | | | | |
| Breastfeeding Professional Peer Support | Participants initiate contact | | Particip | oants atter | nd 2 to 4 s | essions as | needed | |
| Breastfeeding Telephone Assessment (15-20 minutes) | | Χ | Χ | Χ | Х | Χ | Χ | Χ |

**Breastfeeding curriculum.** The Kansas Breastfeeding Coalition, Inc. (KBC) in partnership with the Kansas Department of Health and Environment (KDHE) Bureau of Family Health (Title V

Maternal and Child Health Services Program) created a 2-hour breastfeeding class for parents and parents-to-be. The curriculum aligns with nutritional requirements set by the U.S. Department of Agriculture's Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) and with parenting and maternity care practices of specific Kansas-based organizations such as the Kansas Infant Death and SIDS Network, Inc. 111 and the United Methodist Health Ministry Fund's High 5 for Mom & Baby. 112 Further, the curriculum is based on the Office on Women's Health "Your Guide to Breastfeeding." 113 The content of the 2-hour session will focus on the following areas: establishing and maintain a sufficient and safe breast milk supply, breast anatomy and physiology, maternal diet and lifestyle choices, prescription and non-prescription medications, infant stomach capacity, baby behavior feeding cues, breast milk expression, safe handling and storage of breast milk, returning to work, safe preparation of infant formula, biologically appropriate bottle feeding, and local community breastfeeding resources.

Potential survey participants will have the option of contacting researchers with any questions prior to completing the survey or prior to participating in the educational session, and will self-administer the survey if wanting to participate. Responses will be entered in REDCap for data analysis. All identifying information will be removed from the data prior to analysis. Research personnel will not have access to any identifying information contained in the survey.

Self-Administered Surveys and Incentive to Participate. All surveys will be self-administered (Appendix 1 through 5 – Survey Instruments) and are available in English. The pre- and post-survey instruments are identical. They will be administered electronically at baseline (at study entry) and at six months postpartum (see Table 5 Data Collection). Via email, the study coordinator will provide each participant with a REDCap link that provides electronic access to each survey. Informed consent will occur when the participant opens the survey. Participants will self-administer the survey and may stop at any time. Potential survey participants will have the option of contacting researchers with any questions prior to completing the survey. The survey instrument will be set up using REDCap and responses will be automatically entered and stored in REDCap for data analysis. All identifying information will be removed from the data prior to analysis. Research personnel will not have access to any identifying information contained in the survey.

At recruitment and at study closure 6 months postpartum, <u>all</u> participants will complete four preand post-survey instruments: (1) Breastfeeding assessment, socio-demographic characteristics, and health status (sociodemographic and health status questions will only be asked at baseline, not at study closure) (Appendix 1); (2) Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) (Appendix 1); (3) Kaiser Physical Activity Survey (KPAS) (Appendix 2); (4) the Eating At America's Table Study (EATS) Fruit & Vegetable Intake Screener (Appendix 3) supplemented with questions on fiber, added sugars, dairy, calcium, and meat from the Dietary Screener in the National Health and Nutrition Examination Survey (NHANES 2009-10) (Appendix 4). (Appen

evidence shows that higher BMI pregnant women may have an increased likelihood of postnatal depression. Therefore, at 6 weeks postpartum, all participants will complete the Edinburgh Postnatal Depression Scale (EPDS) (Appendix 5), 127-129 which takes about 5 minutes. Participants with an EPDS score of 10 or higher will be referred to a mental healthcare professional for further psychological evaluation. All study survey instruments are listed in Table 4.

Table 4. Survey Instruments

| Study Instrument | Items Measured | No. of Items | Reliability | Populations Validated |
|---|---|---|---|---|
| Breastfeeding Knowledge Assessment, Socio-<br>demographic Characteristics, and Health Status | To assess knowledge of<br>breastfeeding (44 items), to<br>assess socio-demographic<br>characteristics (6 items), to<br>assess health status (7<br>items) | 57 items; multiple choice,<br>and Likert-type scale | Not yet performed. | Not yet performed. |
| Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | To assess levels of self-<br>efficacy in postpartum<br>women. BSES-SF has also<br>been used with prenatal<br>women. | scale. | Crohnbach's alpha = 0.97 | Postpartum women at 1 week, 4 weeks, and 8 weeks. |
| Kaiser Physical Activity Survey (KPAS) | To assess multiple<br>domains of physical activity<br>and total physical activity in<br>pregnant women. | | Correlation coefficient for total activity: $r = 0.84$ ; correlation coefficient for multiple domains: $r = 0.76 - 0.86$ | Pregnant women aged 18 to<br>47 years old. |
| Fruit & Vegetable Intake Screener (EATS) | To assess intake of fruits and vegetables. | 10 items; with portion-size questions. | Correlation coefficient between test instrument and true intake: $r = 0.51-0.67$ Correlation coefficient between three screeners: $r = 0.52 - 0.71$ | Men and women aged 20 to 70 years old. |
| Selected items from the Dietary Screener<br>Questionnaire (NHANES 2009-10) | To assess intake of fiber,<br>added sugars, dairy,<br>calcium, and meat. | Up to 6 selected items on<br>fiber, added sugars, dairy,<br>calcium and meat; DSQ has<br>a total of 26 items. | Not yet performed. | Not yet performed. |
| Edinburgh Postnatal Depression Scale (EPDS) | To assess levels of depression during the postpartum period. | 10 items | Sensitivity: 34-100%<br>Specificity: 44-100%<br>Positive likelihood ratios: 1.61-78 | Antepartum and postpartum women. |

Each participant will receive a \$50 gift card at consent, after she will deliver her baby, the participant will receive a digital scale and a pedometer, and upon completion of the study (at 6 months after birth), each participant may select a gift up to \$75 for their baby from their baby registry at Walmart. In summary, for participants randomized to any of the three groups: 1) DPP plus breastfeeding, or 2) DPP only, or 3) Usual care, the total possible compensation is valued at \$187.50 including the following gift items: digital scale (valued at \$50 each), pedometer (valued at \$12.50 each), baby gift at Walmart (valued at \$75 each), and a \$50 gift card.

If a participant ends early prior to completing the study, then she will only receive the items for the program components that she completed.

Study payments are taxable income. Prior to distribution of gift items and after obtaining consent, a form 1099 will be provided to each participant for completion. This process is in accordance and in compliance with regulations set forth by the University of Kansas School of Medicine and the Internal Revenue Service if you receive \$600 or more in a calendar year for participating in research studies.

### **Section III. Statistical Methods and Data Analysis**

Study data will be managed using REDCap electronic data capture tools hosted at the University of Kansas School of Medicine – Wichita.<sup>19</sup> REDCap (Research Electronic Data Capture) is a secure, web-based application designed to support data capture for research studies, providing 1) an intuitive interface for validated data entry; 2) audit trails for tracking data manipulation and export procedures; 3) automated export procedures for seamless data downloads to common statistical packages; and 4) procedures for importing data from external sources.

Outcome Measures and Rationale for Outcome Measures. The expected outcomes of this study are (1) to increase postpartum weight loss; (2) to improve HbA1c and mean arterial blood pressure; and (3) to increase any breastfeeding. As this is a pilot trial, we will also collect the following data: number of women screened, number of women recruited and enrolled, number of women who withdraw from the study and reasons for withdrawal, number of women who complete the DPP protocol, and number of women who complete the breastfeeding sessions. Upon recruitment into the study and at study closure, all participants will complete the BSES-SF, KPAS, EATS, and selected items from the DSQ NHANES 2009-10 to assess differences in knowledge and self-efficacy toward breastfeeding, physical activity, and nutrition. Table 5 shows a timeline for data collection in all three study arms.

<u>Aim 1</u>: Test the efficacy of Tx1 to improve 6-month postpartum weight loss among women with a BMI  $\geq$  25. <u>Hypothesis 1</u>: Women in Tx1 will have greater weight loss postpartum compared to women in Tx2 and Tx3. We will measure maternal height and weight as outlined in Table 5 below. We will measure weight loss at the same time points as any breastfeeding because this will allow meaningful comparisons among the study arms.

<u>Aim 2</u>: Test the efficacy of Tx1 to improve 6-month postpartum mean blood glucose (HbA1c) and mean arterial blood pressure among women with a BMI  $\geq$  25. <u>Hypothesis 2</u>: Women in Tx1 will have better HbA1c and mean arterial blood pressure postpartum compared to women in Tx2 and Tx3. We will measure mean blood glucose and mean arterial blood pressure ((systolic blood pressure +2  $^{41}$ /3)) as outlined in Table 5 below. We will also collect baseline data on glucose tolerance levels during pregnancy.

<u>Aim 3</u>: Test the efficacy of Tx1 to increase any breastfeeding through 6 months postpartum among women with a BMI  $\geq$  25. <u>Hypothesis 3</u>: Women in Tx1 will breastfeed longer compared to women in Tx2 and Tx3. At delivery, breastfeeding initiation will be measured (see Table 5). This is defined as starting breastfeeding immediately after delivery. We

will also measure the duration of <u>any</u> breastfeeding (defined as predominant breast milk with some formula supplementation) as outlined in Table 5 below. Further, we will measure exclusivity of breastfeeding (defined as exclusive breast milk without supplementation unless medically necessary), formula supplementation, and solid foods. We will measure formula and solid food at the time that they were first introduced as well as quantity and frequency of feedings.

Table 5. Timeline: Data Collection for All Study Participants

| | Prenatal | | | Postnatal | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Measurements | Baseline | Week 24 | Week 28 | Week 32 | Week 36 | Delivery | 1 Week | 3 Weeks | 6 Weeks | 3 Months | 6 Months |
| Breastfeeding Knowledge, demographics, health status | Χ | | | | | | | | | | Χ |
| Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | Х | | | | | | | | | | Χ |
| Kaiser Physical Activity Survey (KPAS) | Х | | | | | | | | | | Χ |
| Fruit & Vegetable Intake Screener (EATS) | X | | | | | | | | | | Χ |
| Selected items from DSQ (NHANES 2009-10) | Х | | | | | | | | | | Χ |
| Mother's Weight (lbs) | Х | | | | | Χ | Χ | Χ | Χ | Χ | Χ |
| Mother's Height (inches) | Х | | | | | | | | | | |
| Glucose tolerance | Х | | | | | | | | | | |
| Mother's HbA1c | Х | | | | | | | | | | Χ |
| Mother's Mean Arterial Blood Pressure | Х | | | | | Χ | | | | | Χ |
| Baby's Weight (kg) | | | | | | Х | Х | Х | Х | Х | Χ |
| Baby's Height (gm) | | | | | | Х | Х | Х | Х | Х | Χ |
| Breastfeeding Initiation at Delivery | | | | | | Χ | | | | | |
| Breastfeeding Duration (any and exclusive) | | | | | | | Χ | Χ | Χ | Х | Χ |
| Formula Supplementation | | | | | | Х | Χ | Χ | Χ | Χ | Χ |
| Solid Foods | | | | | | | Х | Х | Х | Х | Χ |

Sample Size and Randomization. The primary outcomes of interest are: (1) postpartum weight loss; (2) HbA1c and mean arterial blood pressure; and (3) breastfeeding duration. A total of 60 participants (20 per study arm) will be recruited. The results from this pilot study will be used in sample size estimation for a future study that is sufficiently powered to detect a clinically meaningful effect size. Due to the nature of this project being a feasibility study, the sample size in the proposed study is not based on providing adequate power to detect a clinically meaningful effect size across the three study arms. Block randomization with block size of 5 participants will be employed. A sequence of 12 random integers will be generated using a computer algorithm. The first 4 integers of the sequence will be assigned to the DPP plus breastfeeding arm; the next 4 integers will be assigned to the DPP only arm; and the last 4 will be assigned to the usual care arm. Blocks will be assigned to arms in the increasing order of sequence of integers generated.

**Statistical Analysis.** For baseline data characteristics, descriptive statistics will be reported as mean and standard deviation for continuous variables and as count and percentage for categorical variables. Depending on the distribution of the continuous variables, the Kruskal-Wallis test or ANOVA will be used to test for differences in continuous variables across the three arms. Chi-

Square test of independence (or Fishers exact test if 25% of cells have counts less than 5) will be used to assess the association between categorical variables and the three arms. The analysis will be based on "intention-to-treat" principle. A two-sided alpha level of 0.05 will be used to determine statistical significance. A 95% confidence interval will also be reported.

Aim 1: Test the efficacy of Tx1 to improve 6-month postpartum weight loss among women with a BMI  $\geq$  25. The outcome of interest is 6 month postpartum weight loss measured across the three arms. Weight will be measured at delivery, and at weeks 1, 3, and 6 postpartum and at 3 months (13 weeks) and 6 months (26 weeks) postpartum. The difference in postpartum weight (weight loss) between two consecutive time points will be computed. Thus, each participant has 5 postpartum weight loss values based on weight measurements at 6 different time points. We will use the generalized estimating equation approach to compare weight loss in the DPP plus breastfeeding arm (Tx1) with weight loss in the DPP only (Tx2) and usual care (Tx3) arms, as well as weight loss between Tx2 and Tx3. The working correlation matrix will be specified after assessing the data. The model will be adjusted for the effect of age, race/ethnicity, level of education, annual household income, family history of diabetes, baseline weight, pre-diabetes status, and parity.

Aim 2: Test the efficacy of Tx1 to improve 6-month postpartum mean blood glucose (HbA1c) and mean arterial blood pressure among women with a BMI  $\geq$  25. The outcome of interest is mean blood glucose (HbA1c) and mean arterial blood pressure ((systolic blood pressure +2 (diastolic blood pressure)/3)) measured at baseline, delivery, and at 6 months postpartum across the three arms. We will use a multiple linear regression approach to compare HbA1c in Tx1 with HbA1c in Tx2 and Tx3, as well as HbA1c between Tx2 and Tx3. The model will be adjusted for the effect of age, race/ethnicity, level of education, annual household income, family history of diabetes, pre-diabetes status, parity, and baseline weight. The difference in mean blood arterial pressure at 6 months postpartum will also be assessed using a separate multiple linear regression approach after adjusting for the same covariates listed previously.

Aim 3: Test the efficacy of Tx1 to increase any breastfeeding through 6 months postpartum among women with a BMI  $\geq$  25. The outcome of interest is breastfeeding through 6 months postpartum; it will be measured at delivery, and at weeks 1, 3, and 6 postpartum and at 3 months (13 weeks) and 6 months (26 weeks) postpartum. The risk of stopping "6 month postpartum breastfeeding" in Tx1 relative to Tx2 and Tx3 will be estimated using Zou's modified Poisson regression approach. The outcome in Zou's modified Poisson regression is binary, and it does not take into account the time until which any breastfeeding was done before stopping. However, it provides an interpretation-friendly estimate of the probability of stopping "6 month postpartum breastfeeding." Additionally, the Cox Ph model will be used to compare the risk (hazard) of stopping breastfeeding across each study arm. Unlike Zou's modified Poisson approach, the Cox model takes into account the time of breastfeeding. Any participants who are lost to follow-up will be treated as censored events and participants who stop

breastfeeding during the follow-up are the events of interest. In addition, participants who performed any breastfeeding until 6 months will be treated as administratively censored events. The model will be adjusted for the same covariates listed above under Aims #1 and #2.

Missing data. Owing to the design of the study and non-transient nature of the study population, we anticipate few to none missing observations. Any missing observation that can be attributed to either attrition or nonresponse will be considered missing at random. Depending on the proportion of missingness, complete case analysis (less than 5% missing) or the multiple imputation method will be used to impute missing data. For longitudinal response (postpartum weight measurements), the last observation will be carried forward to impute the missing response. Results based on imputed data will be compared to findings from complete case analysis, to assess the effect of missingness on study findings.

Comparison of scores on the Breastfeeding Assessment, BSES-SF, KPAS, EATS, and selected items from the DSQ. The Breastfeeding Assessment is based on 44 questions. Cronbach's alpha will be used to test the internal consistency of the data. The "difference in Breastfeeding Assessment scores between recruitment and at study closure" across all three study arms will be assessed using the multiple linear regression approach. The model will be adjusted for the effect of age, race/ethnicity, level of education, annual household income, family history of diabetes, pre-diabetes status, and parity. The BSES-SF score is based on 14 questions and ranges from 14 to 70 points. Cronbach's alpha will be used to test the internal consistency of the data. The "difference in BSES scores between recruitment and at study closure" across all three study arms will be assessed using the multiple linear regression approach. The model will be adjusted for the effect of age, race/ethnicity, level of education, annual household income, family history of diabetes, pre-diabetes status, and parity. The KPAS score comprises of 38 questions that are distributed sequentially but non-uniformly across four sections and measure household and family care activities (household index); occupational activities (occupational index); active living habits (active living index); and participation in sports and exercise (sports and exercise index). For each section, Cronbach's alpha will be used to test the internal consistency of the data. For each index of physical activity, "difference/change between recruitment and at study closure" across all three study arms will be assessed using the multiple linear regression approach after adjusting for the effect of the previously stated covariates. The EATS survey consists of 10 questions, and up to 6 questions will be selected from the DSQ. For each question, counts and percentages will be reported for participants at recruitment and at study closure across all three study arms.

#### Section IV. Patient Protections and Methods to Minimize Risk

- A. Risks to Human Subjects
- a. Human Subjects Involvement, Characteristics, and Design

The focus of this research is to implement and determine the feasibility and efficacy of an intervention that is based on the Diabetes Prevention Program (DPP) and includes intensive breastfeeding support and counseling in a cohort of overweight or obese pregnant women to be followed during pregnancy through 6 months postpartum. Study participants will be pregnant women who reside in or near Wichita and in or near Lakin, Kansas. Participants are eligible if they meet study inclusion criteria. This is a randomized controlled pilot study with three study arms. Participants will be randomized to each arm of the study by computer. Participants in Tx1 will receive the DPP plus breastfeeding, participants in Tx2 will receive the DPP only, and participants in Tx3 will receive usual care. Usual care consists of (1) the same obstetrical care that pregnant women with normal body mass index (BMI) receive, and (2) obstetrical care that is provided to pregnant women by the same provider (Dr. Michael Wolfe). Total enrollment for the proposed study will be 60 pregnant female participants.

Participants are recruited from an obstetrical clinic at Via Christi Hospitals Wichita, Inc., a regional medical center located in Wichita, Kansas, and Kearny County Hospital, a critical access full-spectrum rural hospital, in Lakin, Kansas. Participants must be women 18 years old or older, pregnant, with a BMI ≥ 25 and <35, and able to read and understand English. Eligible participants will be recruited during the 1<sup>st</sup> trimester or early during the 2<sup>nd</sup> trimester. General study exclusions include women who have pregnancy complications that require emergency care, have thyroid disease, have multiple gestation, had substance abuse within last 3 years, have an ART (Assisted Reproductive Technology) pregnancy, are a current smoker, had prior bariatric surgery, have been in a weight-loss program within 3 months of conception, have a BMI ≥ 35, are unable to attend intervention/follow-up visits, are unwilling to self-monitor data collection, are unable to complete the intervention, have a presence of any condition that limits walking, have a presence of any condition that limits following diet recommendations, or have a pregnancy complicated with a fetus diagnosed with lethal malformations/conditions.

Vulnerable populations in this study might include economically/educationally disadvantaged persons. Some pregnant women may be economically and/or educationally disadvantaged based on their demographic profile. We especially want to accommodate these individuals as our study's focus is on measuring postpartum weight, breastfeeding behaviors, HbA1c and blood pressure among an at-risk ethnically and racially diverse, overweight and obese pregnant population.

We will obtain approval from the Institutional Review Board (IRB) at the University of Kansas School of Medicine-Wichita (KUSM-W), Via Christi Hospitals Wichita, Inc. (VCH), and Kearny County Hospital (KCH). Via Christi Hospitals Wichita, Inc. and Kearny County Hospital are agreeable to allow Dr. Jacobson and her research team access to use their patient population to recruit study participants. With the active assistance of Dr. Wolfe, maternal fetal medicine specialist at both hospitals, Dr. Jacobson and her research team will recruit each participant for the study. All members of the research team involved in consenting and enrolling participants have successfully completed institutional Human Subjects training.

### b. Sources of materials

Research material obtained from participants will include: socio-demographic data (i.e. age, race/ethnicity, income, education level, etc.), breastfeeding self-efficacy, physical activity level, dietary assessment, level of postpartum depression, weight, height, HbA1c, mean arterial blood pressure, blood glucose tolerance level during pregnancy, breastfeeding initiation, breastfeeding duration, use of formula, and solid food. All data are based on validated questionnaires (except for the Breastfeeding Assessment questionnaire), and activity and nutrition monitoring as required by the DPP protocol. The validated measures that will be used are the Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), the Kaiser Physical Activity Survey (KPAS), the Fruit and Vegetable Intake Screener (EATS), the Dietary Screener Questionnaire (NHANES 2009-10), and the Edinburgh Postnatal Depression Scale (EDPS). These validated survey instruments will be administered at baseline (=study entry) and at study closure (=6 months postpartum). At delivery and through the 6 month postpartum period, we will also obtain the infant's height and weight. Further, at delivery, we will measure if the mother will start breastfeeding and we will measure how long she will continue breastfeeding through 6 months postpartum.

All behavioral assessments/surveys will be completed in a private room without the researcher present. All DPP orientation sessions and breastfeeding classes will take place at Via Christi Health or Kearny County Hospital (depending on the residence of the study participant). Data collected will be stored on a secure drive backed up on a nightly basis by the Information Technology (IT) department at KUSM-W. Identification numbers will be assigned to each participant at the time of initial survey completion. All hard-copy and data files will be labelled according to participant number. Only the research team will have access to information regarding demographic and medical information and identification number for each participant. All other data collected throughout the duration of the study will be kept in locked cabinets and on a secure server within the University of Kansas School of Medicine-Wichita. Data used for analysis will be de-identified and accessible only by the research team. A log will be kept of all data collection and analysis steps completed for each participant.

### c. Potential risks

Participants will undergo an intervention that is educational. Participants will share education on exercise and diet, and will then apply these concepts in their daily functioning. During the study, participants' weight, HbA1c and mean arterial blood pressure will be measured. During pregnancy, the breastfeeding component of the proposed intervention is highly visual and interactive. An International Board Certified Lactation Consultant (IBCLC) will demonstrate proper breastfeeding techniques and strategies. After delivery, participants will have access to an IBCLC up to 6 months postpartum. There are no known risks of subjects participating in an educational intervention. All data will be kept anonymous and in a locked file cabinet in a locked office. All data will be entered into a computer; electronic data will be on a secure server at KUSM-W that is backed up on a nightly basis by the IT department at KUSM-W.

A potential risk of participating in the study is a breach of confidentiality and loss of privacy. Privacy measures for participant responses to the questionnaires are described below. Yet, to further address privacy, as well as to insure confidentiality, the investigators will ensure the following measures are taken. All data obtained in the study will be kept confidential. The only parties having access to the data in the proposed study will be the Principal Investigator (Dr. Jacobson), Dr. Jacobson's research team, and the Institutional Review Board of record. Hardcopies of completed participant questionnaires will be locked in a secure file cabinet in the PI's office. Responses to the surveys and the clinical information obtained will be maintained on the KUSM-W REDCap database. Only the necessary members of the research team will have access to the REDCap database.

# **B.** Adequacy of Protection Against Risks

### a. Recruitment and Informed Consent

Participants will be recruited from the obstetrical clinic located at Via Christi Hospitals Wichita, Inc., a regional medical center located in Wichita, Kansas, and at Kearny County Hospital, a critical access full-spectrum rural hospital, in Lakin, Kansas. We will use printed flyers, posters and word-of-mouth advertising to recruit potential participants. Prior to using these recruitment materials, IRB at Via Christi Hospitals Wichita, Inc. will review and approve these materials. Dr. Michael Wolfe, Via Christi Hospitals Wichita, Inc. and Kearny County Hospital's maternal fetal medicine specialist, will make the initial contact with a potential participant during her first prenatal visit and screen for inclusion criteria. If Dr. Wolfe believes a potential participant meets inclusion criteria, then he will familiarize her with the nature and purpose of the study. If the potential participant is interested in the study, then he will give her a study brochure and a hard paper copy of the consent form. Prior to using this study brochure, the brochure will be reviewed and approved by the IRB at Via Christi Hospitals Wichita, Inc. By providing the potential participant with a copy of the consent form, this will serve as the verbal consent script.

Then, Dr. Wolfe will provide Dr. Jacobson and her research coordinator the potential participant's contact information (i.e., participant name, email address, telephone number). After receiving a potential participant's name and phone number from Dr. Wolfe, the research coordinator will follow up with a phone call or meet with the interested participant in-person in an on-site, private conference room immediately after their prenatal appointment to determine if the potential participant again meets study inclusion criteria. If she does, the coordinator will screen if the potential participant meets study exclusion criteria during the same phone call or during this same in-person on-site visit (see Table 1). Before the research coordinator screens for inclusion and exclusion criteria, during this same phone call or during this same in-person on-site visit, verbal consent will be obtained between the participant and the research coordinator, using the consent form as the verbal consent script, and then written e-consent will be obtained via REDCap at the orientation session. When a participant is recruited on-site, then the in-person visit between the participant and the research coordinator is considered to be the orientation session.

If the participant meets all study criteria and the participant is contacted via telephone and not inperson on-site, then the research coordinator will provide her with a time and place for the DPP's orientation session and to complete study-related survey instruments. The research coordinator will also verify the participant's email address to provide her with informed consent materials for review. Study procedures will be explained verbally by the PI and in writing at the time of survey completion and, again, at the DPP's orientation session. All subjects participating in the study will consent to participate as evidenced by signing an informed e-consent form via REDCap immediately prior to commencement of the orientation session. Subjects will be informed that they are free to withdraw their consent at any time during the study with no penalty.

Written informed e-consent will be obtained via REDCap from each participant prior to completing the first questionnaire. A verbal explanation of the study will be provided in addition to the written explanation included in the consent form. Potential participants will be encouraged to ask questions concerning the study. After reading the consent form, participants will be asked to provide a verbal summary of the study as they understand it. This will be used to assess the participant's understanding of the study. If potential participants are able to understand, remember, and verbalize the main aspects of the study, it will be assumed that they have the capacity to consent. Participants will be informed that they can withdraw from the study at any time by contacting research personnel. When consent is withdrawn, participation in the study will be terminated and no additional data will be collected or used for analysis. All patients will receive a copy of their signed consent form. The original signed consent forms will be kept in a locked file cabinet in a secure data storage room in Dr. Jacobson's office area, which can only be accessed with a key.

#### b. Protection Against Risk

All information we obtain throughout the study will be kept confidential. The risks associated with the study are minimal. No adverse events are anticipated with this study, but procedures will be in place to monitor the study using the scientific protocol provided and approved by the Institutional Review Board of record. Participants experiencing any adverse effects from participating in this study will be directed to the PI. Action will be taken to direct the study participant to the appropriate resources.

Information collected throughout the course of the study will be de-identified of Protected Health Information (PHI), and will only be accessed by research staff directly involved with the study. Researchers believe there is less than minimal risk regarding economic risks and legal risks pertaining to this study. However, the risks associated with this project are considerably reasonable in comparison to the potential benefits from the study.

### c. Adverse Events

In the case an adverse event were to occur due to study procedures, the principal investigator, Dr. Jacobson, will assume responsibility for reporting and documenting any complications. All adverse events will be recorded and the necessary documents will be completed. The principal investigator and/or the project coordinator will notify the IRB within the appropriate time frame. The investigators and project coordinator are responsible for complying with any reporting requirement of the reviewing IRB.

If an adverse event should occur, the participant will have the opportunity to withdraw from the study. Dr. Wolfe will be available for consultation should an adverse event happen. Throughout the study, we will be monitoring for issues related to safety of participants as well as privacy of data. Should an adverse event occur, the research team will document the event. The following information will be monitored throughout the study: number of participants screened and enrolled, drop-outs, and serious and non-serious adverse events. This data, with the exception of serious adverse events, will be reported every 12-months. Because no serious adverse events are anticipated in this study, any such events will be immediately reported to the Institutional Review Board of record. If the severity of an adverse event requires emergency medical attention, appropriate providers/staff will be contacted to provide medical attention. To assess participant safety even further, we will have a Data and Safety Officer in place. Dr. Paige Geiger has agreed and is confirmed as the Data and Safety Officer for our study. Paige Geiger, PhD, is a full professor in the Department of Molecular and Integrative Physiology, University of Kansas School of Medicine-Kansas City, Mailstop 3043, 3901 Rainbow Boulevard, Kansas City, KS 66160.

### C. Potential Benefits of the Proposed Research to the Subjects and Others

The potential benefit of this study is to determine if a combined breastfeeding, DPP-based intervention reduces postpartum weight, increases breastfeeding, and improves mean blood glucose (HbA1c) and mean arterial blood pressure, among an at-risk population with a BMI ≥ 25. This is an innovative way to address physical activity, weight, and breastfeeding in one intervention that is modeled after the evidence-based Diabetes Prevention Program and could be integrated into the continuum of healthcare services provided to culturally, diverse at-risk pregnant women. Results of the proposed intervention will inform the development of interventions aimed at reducing diabetes risk factors and potential progression to type 2 diabetes after pregnancy among at-risk women. The overall impact of this project will be to reduce diabetes risk factors among a high-risk population and inform interventions aimed at reducing these risk factors thereby decreasing disproportionate morbidity. Moreover, study results will add significant knowledge to the field of diabetes prevention and related behavioral health interventions and strategies to improve maternal and child health outcomes. Although the randomization process will not be performed by a clinician, instead it will be generated by a computer system, participants may still have concerns about bias (who receives the treatment versus who receives the control). We will inform them that, regardless of group assignment, they will continue to receive routine care from their maternal fetal medicine specialist.

### D. Importance of the Knowledge to be Gained

Knowledge to be gained from this study is whether a combined breastfeeding, DPP-based intervention reduces diabetes risk factors among an at-risk population. Results of this study will enhance current intervention efforts that aim to reduce diabetes risk factors and potential progression to diabetes during and after pregnancy and improve breastfeeding thereby improving maternal and child health outcomes. An intervention that starts during pregnancy and extends beyond pregnancy has a high likelihood of success because during this time period, women are more inclined to change their behavior to benefit their children leading to reduced risk of retaining excess weight and a possible subsequent healthier pregnancy. The knowledge, methodologies, and strategies obtained from this study will be of importance to the submission of a larger research grant such as an R01with the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) that will involve a longitudinal study with a larger sample size of high-risk, ethnically and racially diverse Kansas women and their children to assess if a combined breastfeeding, DPP-based program reduces maternal risk for diabetes and impedes the cycle of obesity as a diabetes risk factor among families. The R01 is a Research Project Grant and is the original and historically oldest grant mechanism used by the National Institutes of Health (NIH). The R01 provides support for health-related research and development based on the mission of the NIH. An R01 can be investigator-initiated or can be solicited via a Request for Applications by the NIH. The R01 is an award made to support a discrete, specified, circumscribed project to be performed by the named investigators in an area representing the investigators' specific interest and competencies, based on the mission of the NIH. It is believed that the minimal risk involved in the proposed study is reasonable considering that it could lead to more effective ways to reduce diabetes risk factors among at-risk populations with a greater burden of disease and risk for related health complications. The proposed pilot study will be the first to use an intensive breastfeeding, DPP-based program to reduce diabetes risk factors among a vulnerable, at-risk population.

### E. Privacy and Confidentiality

This is an educational intervention utilizing identified pre- and post-surveys. The privacy and confidentiality of potential participants will be maintained as all study data will be protected and only study personnel have access.

Only the listed investigators and their designated staff will have access to the surveys and study data. The University of Kansas School of Medicine-Wichita IRB, the US Department of Health and Human Services, the Office of Human Research Protections, and other government and regulatory bodies as required by law may have access to these research data. Information technology protections and firewalls are in place at all study facilities, and will protect the electronic data stored at each facility. Secure email will be used to transfer documents between investigators. The database (participant identifiers removed) will be encrypted and password-protected when sent through secure email between investigators.

### F. Waiver of Documentation of Consent

A Waiver of Documentation of Consent is <u>not</u> requested for this study. This study presents no more than minimal risk to study participants as the information obtained is not sensitive in nature, and if inadvertently released should not be injurious to the participants, either financially, legally, or personally. Surveys will not ask for a participant's name, medical record number, birthdate, social security number, or any other protected health information. However, it is critical that the pre- and post-surveys, along with data on individual weight loss, HbA1c, mean arterial blood pressure and length of breastfeeding are linked to the same individual to assess health outcomes. Therefore, research personnel will seek informed written consent and the process for obtaining written consent is outlined previously under <u>Item B</u>. Adequacy of Protection Against Risks, Item a. Recruitment and Informed Consent.

### G. Adherence to Study Protocol

Protocol adherence is the primary responsibility of the principal investigator. The co-investigators will serve to support protocol adherence efforts and maintain an understanding of all protocol details. Protocol amendments, revisions, deviations will be promptly reported to the IRB.

### H. Secure and Maintain IRB Approval at All Sites

IRB approval will include all the study locations listed previously. All protocol deviations, amendments, revisions, and continuing review reports will be promptly compiled and reviewed by the principal investigator and co-investigators, and provided to the IRB. All research within the scope of this project will be conducted under IRB policies and guidelines.

# I. Obtain IRB Approvals Prior to Implementing Changes to Protocol

The principal investigator and co-investigators wish to assure the IRB that any amendments to the protocol or supporting documents will be submitted for approval prior to implementation; problems associated with the research will be reported in accordance with IRB policies.

# J. Modifications to Study Protocol and Oversight

Each review will consider whether or not the study should continue without change, be modified, or be terminated. Recommendations regarding modification of the design and conduct of the study might include:

- 1. Modification of the study protocol based upon review of the safety data;
- 2. Optional approaches when the incidence of primary study outcomes is substantially less than expected such as recommendations to extend study site;
- 3. Corrective actions regarding the study site.
- 4. To assess participant safety, we will have a Data and Safety Officer in place.

The principal investigator and co-investigators will provide oversight, supervision and monitoring of the data collection and will insure integrity of the data which will ultimately ensure subject confidentiality.

### **K.** Monitoring Unanticipated Problems

The principal investigator, Lisette Jacobson, will assume responsibility for:

- 1. Data quality, completeness, and timeliness;
- 2. Adherence to the protocol;
- 3. Factors that might affect the study outcome or compromise the confidentiality of the trial data (such as protocol deviations).

The principal investigator will consult with the research team/co-investigators regarding protocol revisions and amendments before adopting such changes. The IRB will be notified of any problems during the conduct of this study.

### L. Ensure General Coordination of Study Conduct

The principal investigator agrees to accept responsibility for the scientific conduct of this study and for the rights and welfare of human subjects. General oversight of the coordination of this study will be provided by the principal investigator.

#### M. Record Retention

All other study related documents (protocols, databases, IRB documents, surveys) will be retained for fifteen (15) years from the data of initial IRB approval and will be kept in the principal investigator's office (University of Kansas School of Medicine - Wichita) under lock and key at the conclusion of this study. At the time of document disposal, documents will be shredded according to KUMC Research Institute Record Retention guidelines. The University of Kansas School of Medicine record retention policy requires research records involving human subjects to be kept for at least 15 years so all data associated with this study will be kept for at least 15 years.

### Section V. Results, Source of Funding, and Study Timeline

#### A. Dissemination of Results

The findings of this study will be submitted to peer reviewed public health and diabetes prevention journals (i.e. American Journal of Public Health, Diabetes, Diabetes Care, Diabetes Obesity and Metabolism, Health Education and Behavior, Maternal Child Health Journal, etc.), and may be presented at conferences (i.e. Society of Behavioral Medicine, American Public Health Association, American Diabetes Association, National Rural Health Association, research forums, ACOG, district meetings, obstetrical updates, etc.). The IRB will be notified at time of continuing review of the research project. Additionally, findings will be used in the future to obtain grant funding and for future intervention development.

#### **B.** Source of Funding

This study will be funded by the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), grant number 1K01DK113048-01A1.

### C. Study Timeline (tentative)

The following timeline is suggested for study completion.

| Suggested Timeframe | Completed Objective/Goals |
|---|---|
| September 2018 – December 2018 | IRB protocols, preliminary work including |
| | hiring of research coordinator, and working |
| | working with clinical staff at both hospital |
| | sites |
| January 2019 – August 2019 | Finalize planning for participant |
| | recruitment |
| September 2019 | Start recruitment (rolling recruitment over a |
| | 9 month period) |
| September 2019 – September 2021 | Intervention, data collection, preliminary |
| | data analysis |
| September 2021 | Intervention/trial closes |
| September 2021 – December 2022 | Final data analysis, manuscript completion, |
| | dissemination of findings, preparation for |
| | R01 submission |
| January 2023 – September 2023 | R01 submission |

### **Section VI. Attachments/Appendices:**

- 1. Appendix 1 Survey Instrument, Breastfeeding Self-Efficacy Scale-Short From (BSES-SF) and Breastfeeding Knowledge Assessment (the Breastfeeding Knowledge assessment includes questions regarding socio-demographic data and health status data; these data will only be collected at study entry)
- 2. Appendix 2 Survey Instrument, Kaiser Physical Activity Survey (KPAS)
- 3. Appendix 3 Survey Instrument, Eating at America's Table Study (EATS) Fruit and Vegetable Intake Screener
- 4. Appendix 4 Selected survey items (6) from the "Dietary Screener Questionnaire" (NHANES 2009-10)
- 5. Appendix 5 Survey Instrument, Edinburgh Postnatal Depression Scale (EPDS)
- 6. Appendix 6 Bristol Breastfeeding Assessment Tool (BBAT)
- 7. Appendix 7 Letter of Support from Via Christi
- 8. Appendix 8 Letter of Support from Kearny County Hospital
- 9. Appendix 9 Letter of Support from Dr. Michael Wolfe

### References

- 1. Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. *American journal of obstetrics and gynecology.* 1982;144(7):768-773.
- 2. DeSisto CL, Kim SY, Sharma AJ. Prevalence Estimates of Gestational Diabetes Mellitus in the United States, Pregnancy Risk Assessment Monitoring System (PRAMS), 2007-2010. *Preventing Chronic Disease*. 2014;11:E104.
- 3. Classification and diagnosis of diabetes mellitus and other categories of glucose intolerance. National Diabetes Data Group. *Diabetes*. 1979;28(12):1039-1057.
- 4. Metzger BE, Gabbe SG, Persson B, et al. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. *Diabetes care*. 2010;33(3):676-682.
- 5. Chen P, Wang S, Ji J, et al. Risk factors and management of gestational diabetes. *Cell Biochem Biophys.* 2015;71(2):689-694.
- 6. Cypryk K, Szymczak W, Czupryniak L, Sobczak M, Lewinski A. Gestational diabetes mellitus an analysis of risk factors. *Endokrynol Pol.* 2008;59(5):393-397.
- 7. Bottalico JN. Recurrent gestational diabetes: risk factors, diagnosis, management, and implications. *Seminars in perinatology*. 2007;31(3):176-184.
- 8. Mao L, Ge X, Xu Y, et al. [Pregestational body mass index, weight gain during first half of pregnancy and gestational diabetes mellitus: a prospective cohort study]. *Zhonghua Liu Xing Bing Xue Za Zhi.* 2015;36(5):416-420.
- 9. Spong CY, Guillermo L, Kuboshige J, Cabalum T. Recurrence of gestational diabetes mellitus: identification of risk factors. *Am J Perinatol.* 1998;15(1):29-33.
- 10. Council IoMaNR. Weight gain during pregnancy: Reexamining the guidelines. 2009: http://www.nap.edu/openbook.php?record\_id=12584.
- 11. Gunderson EP, Abrams B, Selvin S. The relative importance of gestational gain and maternal characteristics associated with the risk of becoming overweight after pregnancy. *International journal of obesity and related metabolic disorders : journal of the International Association for the Study of Obesity.* 2000;24(12):1660-1668.
- 12. Oken E, Taveras EM, Kleinman KP, Rich-Edwards JW, Gillman MW. Gestational weight gain and child adiposity at age 3 years. *American journal of obstetrics and gynecology*. 2007;196(4):322 e321-328.
- 13. Siega-Riz AM, Viswanathan M, Moos MK, et al. A systematic review of outcomes of maternal weight gain according to the Institute of Medicine recommendations: Birthweight, fetal growth, and postpartum weight retention. *American journal of obstetrics and gynecology.* 2009;201(4):339 e331-314.
- 14. Stotland NE, Cheng YW, Hopkins LM, Caughey AB. Gestational weight gain and adverse neonatal outcome among term infants. *Obstetrics and gynecology.* 2006;108(3 Pt 1):635-643.
- 15. Al-Kubaisy W, Al-Rubaey M, Al-Naggar RA, Karim B, Mohd Noor NA. Maternal obesity and its relation with the cesarean section: a hospital based cross sectional study in Iraq. *BMC pregnancy and childbirth.* 2014;14:235.

- 16. Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. *Lancet*. 2009;373(9677):1773-1779.
- 17. Lee AJ, Hiscock RJ, Wein P, Walker SP, Permezel M. Gestational diabetes mellitus: clinical predictors and long-term risk of developing type 2 diabetes: a retrospective cohort study using survival analysis. *Diabetes care*. 2007;30(4):878-883.
- 18. Ovesen PG, Jensen DM, Damm P, Rasmussen S, Kesmodel US. Maternal and neonatal outcomes in pregnancies complicated by gestational diabetes. a nation-wide study. *The journal of maternal-fetal & neonatal medicine : the official journal of the European Association of Perinatal Medicine, the Federation of Asia and Oceania Perinatal Societies, the International Society of Perinatal Obstet.* 2015:1-5.
- 19. Saydah SH, Chandra A, Eberhardt MS. Pregnancy experience among women with and without gestational diabetes in the U.S., 1995 National Survey Of Family Growth. *Diabetes care*. 2005;28(5):1035-1040.
- 20. Metzger BE, Lowe LP, Dyer AR, et al. Hyperglycemia and adverse pregnancy outcomes. *N Engl J Med.* 2008;358(19):1991-2002.
- 21. Yogev, Chen, Hod, et al. Hyperglycemia and Adverse Pregnancy Outcome (HAPO) study: preeclampsia. *American journal of obstetrics and gynecology.* 2010;202(3):255 e251-257.
- 22. Catalano PM, McIntyre HD, Cruickshank JK, et al. The hyperglycemia and adverse pregnancy outcome study: associations of GDM and obesity with pregnancy outcomes. *Diabetes care*. 2012;35(4):780-786.
- 23. Srichumchit S, Luewan S, Tongsong T. Outcomes of pregnancy with gestational diabetes mellitus. *International journal of gynaecology and obstetrics: the official organ of the International Federation of Gynaecology and Obstetrics.* 2015;131(3):251-254.
- 24. Young BC, Ecker JL. Fetal macrosomia and shoulder dystocia in women with gestational diabetes: risks amenable to treatment? *Current diabetes reports*. 2013;13(1):12-18.
- 25. Shefali AK, Kavitha M, Deepa R, Mohan V. Pregnancy outcomes in pre-gestational and gestational diabetic women in comparison to non-diabetic women--A prospective study in Asian Indian mothers (CURES-35). *The Journal of the Association of Physicians of India.* 2006;54:613-618.
- 26. Mitanchez D, Yzydorczyk C, Siddeek B, Boubred F, Benahmed M, Simeoni U. The offspring of the diabetic mother Short- and long-term implications. *Best practice & research Clinical obstetrics & gynaecology.* 2015;29(2):256-269.
- 27. ACOG Practice Bulletin No. 22: Fetal Macrosomia. *Obstetrics and gynecology*. 2013;96(5).
- 28. Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. *Obstetrics and gynecology*. 2013;122(5):1122-1131.
- 29. Gonen O, Rosen DJ, Dolfin Z, Tepper R, Markov S, Fejgin MD. Induction of labor versus expectant management in macrosomia: a randomized study. *Obstetrics and gynecology*. 1997;89(6):913-917.
- 30. ACOG Committee Opinion No. 586: Health disparities in rural women. *Obstetrics and gynecology*. 2014;123(2 Pt 1):384-388.

- 31. Chandler D. Late entry into prenatal care in a rural setting. *The Journal of Midwifery & Women's Health*. 2002;47(1):28-34.
- 32. Gallagher A, Liu J, Probst JC, Martin AB, Hall JW. Maternal obesity and gestational weight gain in rural versus urban dwelling women in South Carolina. *The Journal of rural health: official journal of the American Rural Health Association and the National Rural Health Care Association.* 2013;29(1):1-11.
- 33. Rayburn WF, Richards ME, Elwell EC. Drive times to hospitals with perinatal care in the United States. *Obstetrics and gynecology.* 2012;119(3):611-616.
- 34. Strutz KL, Dozier AM, van Wijngaarden E, Glantz JC. Birth outcomes across three rural-urban typologies in the Finger Lakes region of New York. *The Journal of rural health : official journal of the American Rural Health Association and the National Rural Health Care Association*. 2012;28(2):162-173.
- 35. McElroy JA, Bloom T, Moore K, Geden B, Everett K, Bullock LF. Perinatal mortality and adverse pregnancy outcomes in a low-income rural population of women who smoke. *Birth defects research Part A, Clinical and molecular teratology.* 2012;94(4):223-229.
- 36. Blumenshine P, Egerter S, Barclay CJ, Cubbin C, Braveman PA. Socioeconomic disparities in adverse birth outcomes: a systematic review. *American journal of preventive medicine*. 2010;39(3):263-272.
- 37. Jacobson LT, Twumasi-Ankrah P, Redmond ML, et al. Characteristics associated with breastfeeding behaviors among urban versus rural women enrolled in the Kansas WIC program. *Maternal and child health journal*. 2015;19(4):828-839.
- 38. Jacobson LT, Duong, J., Grainger, D. A., Collins, T. C., Farley, D., Wolfe, M., Dong, F., Anderson, B. Health assessment of a rural obstetrical population in a Midwestern state. *Journal of Pregnancy and Child Health*. 2016;3(2).
- 39. ACOG Practice Bulletin No. 22: Fetal Macrosomia. *Obstetrics and gynecology.* 2013;96(5).
- 40. Metzger BE, Persson B, Lowe LP, et al. Hyperglycemia and adverse pregnancy outcome study: neonatal glycemia. *Pediatrics*. 2010;126(6):e1545-1552.
- 41. Boney CM, Verma A, Tucker R, Vohr BR. Metabolic syndrome in childhood: association with birth weight, maternal obesity, and gestational diabetes mellitus. *Pediatrics*. 2005;115(3):e290-296.
- 42. Mitanchez D, Yzydorczyk C, Siddeek B, Boubred F, Benahmed M, Simeoni U. The offspring of the diabetic mother Short- and long-term implications. *Best practice & research Clinical obstetrics & gynaecology.* 2014.
- 43. Flores G, Lin H. Factors predicting overweight in US kindergartners. *The American journal of clinical nutrition*. 2013;97(6):1178-1187.
- 44. Page KA, Romero A, Buchanan TA, Xiang AH. Gestational diabetes mellitus, maternal obesity, and adiposity in offspring. *The Journal of pediatrics*. 2014;164(4):807-810.
- 45. Nehring I, Chmitorz A, Reulen H, von Kries R, Ensenauer R. Gestational diabetes predicts the risk of childhood overweight and abdominal circumference independent of maternal obesity. *Diabetic medicine : a journal of the British Diabetic Association*. 2013;30(12):1449-1456.

- 46. Freeman J, Ferrer RL, Greiner KA. Viewpoint: Developing a physician workforce for America's disadvantaged. *Academic medicine : journal of the Association of American Medical Colleges.* 2007;82(2):133-138.
- 47. Ross R. Fifteen-year outcomes of a rural residency: aligning policy with national needs. *Fam Med.* 2013;45(2):122-127.
- 48. Gamm LD, Hutchison LL, Dabney BJ, Dorsey AM. *Rural Healthy People 2010: A Companion Document to Healthy People 2010. Volume 1.* College Station, Texas: The Texas A&M University System Health Science Center, School of Rural Public Health, Southwest Rural Health Research Center; 2003.
- 49. Bellamy GR, Bolin JN, Gamm LD. Rural Healthy People 2010, 2020, and beyond: the need goes on. *Family & community health*. 2011;34(2):182-188.
- 50. Allen W. Obstetric care in a rural family practice. *The Journal of the American Board of Family Practice / American Board of Family Practice*. 1989;2(1):30-33.
- 51. Norris TE, Reese JW, Pirani MJ, Rosenblatt RA. Are rural family physicians comfortable performing cesarean sections? *The Journal of family practice*. 1996;43(5):455-460.
- 52. Jacobson LT, Dong F, Scheuermann TS, Redmond ML, Collins TC. Smoking Behaviors Among Urban and Rural Pregnant Women Enrolled in the Kansas WIC Program. *Journal of community health*. 2015.
- 53. Gillman MW, Ludwig DS. How early should obesity prevention start? *N Engl J Med.* 2013;369(23):2173-2175.
- 54. Horan MK, McGowan CA, Gibney ER, Donnelly JM, McAuliffe FM. Maternal diet and weight at 3 months postpartum following a pregnancy intervention with a low glycaemic index diet: results from the ROLO randomised control trial. *Nutrients*. 2014;6(7):2946-2955.
- 55. U.S. Department of Health and Human Services. National Institutes of Health. Diabetes Prevention Program. 2008.
- 56. Ferrara A, Hedderson MM, Albright CL, et al. A pregnancy and postpartum lifestyle intervention in women with gestational diabetes mellitus reduces diabetes risk factors: a feasibility randomized control trial. *Diabetes care*. 2011;34(7):1519-1525.
- 57. Nicklas JM, Zera CA, England LJ, et al. A web-based lifestyle intervention for women with recent gestational diabetes mellitus: a randomized controlled trial. *Obstetrics and gynecology*. 2014;124(3):563-570.
- 58. Gunderson EP, Hurston SR, Ning X, et al. Lactation and Progression to Type 2 Diabetes Mellitus After Gestational Diabetes Mellitus: A Prospective Cohort Study. *Annals of internal medicine*. 2015;163(12):889-898.
- 59. Gunderson EP, Hedderson MM, Chiang V, et al. Lactation intensity and postpartum maternal glucose tolerance and insulin resistance in women with recent GDM: the SWIFT cohort. *Diabetes care*. 2012;35(1):50-56.
- 60. Chouinard-Castonguay S, Weisnagel SJ, Tchernof A, Robitaille J. Relationship between lactation duration and insulin and glucose response among women with prior gestational diabetes. *European journal of endocrinology / European Federation of Endocrine Societies*. 2013;168(4):515-523.

- 61. O'Reilly M, Avalos G, Dennedy MC, O'Sullivan EP, Dunne FP. Breast-feeding is associated with reduced postpartum maternal glucose intolerance after gestational diabetes. *Irish medical journal*. 2012;105(5 Suppl):31-36.
- 62. Binns C, Lee M, Low WY. The Long-Term Public Health Benefits of Breastfeeding. *Asia Pac J Public Health*. 2016;28(1):7-14.
- 63. Kirkegaard H, Stovring H, Rasmussen KM, Abrams B, Sorensen TI, Nohr EA. How do pregnancy-related weight changes and breastfeeding relate to maternal weight and BMI-adjusted waist circumference 7 y after delivery? Results from a path analysis. *The American journal of clinical nutrition*. 2014;99(2):312-319.
- 64. Martin J, MacDonald-Wicks L, Hure A, Smith R, Collins CE. Reducing postpartum weight retention and improving breastfeeding outcomes in overweight women: a pilot randomised controlled trial. *Nutrients*. 2015;7(3):1464-1479.
- 65. Stuebe AM, Rich-Edwards JW. The reset hypothesis: lactation and maternal metabolism. *American journal of perinatology.* 2009;26(1):81-88.
- 66. Bernier MO, Plu-Bureau G, Bossard N, Ayzac L, Thalabard JC. Breastfeeding and risk of breast cancer: A meta-analysis of published studies. *Hum Reprod Update*. 2000;6(4):374-386.
- 67. Danforth KN, Tworoger SS, Hecht JL, Rosner BA, Colditz GA, Hankinson SE. Breastfeeding and risk of ovarian cancer in two prospective cohorts. *Cancer Causes Control*. 2007;18(5):517-523.
- 68. Jordan SJ, Cushing-Haugen KL, Wicklund KG, Doherty JA, Rossing MA. Breast-feeding and risk of epithelial ovarian cancer. *Cancer Causes Control.* 2012;23(6):919-927.
- 69. Stuebe AM, Rich-Edwards JW, Willett WC, Manson JE, Michels KB. Duration of lactation and incidence of type 2 diabetes. *JAMA*. 2005;294(20):2601-2610.
- 70. Schwarz EB, Brown JS, Creasman JM, et al. Lactation and maternal risk of type 2 diabetes: a population-based study. *Am J Med.* 2010;123(9):863 e861-866.
- 71. American Academy of Pediatrics. Breastfeeding and the use of human milk. *Pediatrics*. 2012;129(3):e827-841.
- 72. Saadeh MR. A new global strategy for infant and young child feeding. *Forum Nutr.* 2003;56:236-238.
- 73. Kansas Department of Health and Environment BoFH. Personal communication via electronic mail. 2017.
- 74. Breastfeeding Report Card United States, 2016. <a href="http://www.cdc.gov/breastfeeding/data/reportcard.htm">http://www.cdc.gov/breastfeeding/data/reportcard.htm</a>. Accessed October 1, 2016.
- 75. Scheuermann TS, Richter KP, Jacobson LT, Shireman TI. Medicaid Coverage of Smoking Cessation Counseling and Medication is Underutilized for Pregnant Women. *Nicotine & tobacco research : official journal of the Society for Research on Nicotine and Tobacco.* 2017 (forthcoming).
- 76. Athukorala C, Rumbold AR, Willson KJ, Crowther CA. The risk of adverse pregnancy outcomes in women who are overweight or obese. *BMC pregnancy and childbirth*. 2010;10:56.
- 77. Burstein E, Levy A, Mazor M, Wiznitzer A, Sheiner E. Pregnancy outcome among obese women: a prospective study. *American journal of perinatology*. 2008;25(9):561-566.

- 78. Denison FC, Norwood P, Bhattacharya S, et al. Association between maternal body mass index during pregnancy, short-term morbidity, and increased health service costs: a population-based study. *BJOG*: an international journal of obstetrics and gynaecology. 2014;121(1):72-81; discussion 82.
- 79. Gaillard R, Durmus B, Hofman A, Mackenbach JP, Steegers EA, Jaddoe VW. Risk factors and outcomes of maternal obesity and excessive weight gain during pregnancy. *Obesity (Silver Spring, Md)*. 2013;21(5):1046-1055.
- 80. Bhattacharya S, Campbell DM, Liston WA, Bhattacharya S. Effect of Body Mass Index on pregnancy outcomes in nulliparous women delivering singleton babies. *BMC Public Health*. 2007;7:168.
- 81. Gaillard R, Steegers EA, Duijts L, et al. Childhood cardiometabolic outcomes of maternal obesity during pregnancy: the Generation R Study. *Hypertension*. 2014;63(4):683-691.
- 82. Harpsoe MC, Basit S, Bager P, et al. Maternal obesity, gestational weight gain, and risk of asthma and atopic disease in offspring: a study within the Danish National Birth Cohort. *The Journal of allergy and clinical immunology*. 2013;131(4):1033-1040.
- 83. Hinkle SN, Sharma AJ, Swan DW, Schieve LA, Ramakrishnan U, Stein AD. Excess gestational weight gain is associated with child adiposity among mothers with normal and overweight prepregnancy weight status. *The Journal of nutrition*. 2012;142(10):1851-1858.
- 84. Masho SW, Cha S, Morris MR. Prepregnancy obesity and breastfeeding noninitiation in the United States: an examination of racial and ethnic differences. *Breastfeeding medicine*: the official journal of the Academy of Breastfeeding Medicine. 2015;10(5):253-262.
- 85. Reynolds RM, Allan KM, Raja EA, et al. Maternal obesity during pregnancy and premature mortality from cardiovascular event in adult offspring: follow-up of 1 323 275 person years. *BMJ (Clinical research ed)*. 2013;347:f4539.
- 86. Stothard KJ, Tennant PW, Bell R, Rankin J. Maternal overweight and obesity and the risk of congenital anomalies: a systematic review and meta-analysis. *Jama*. 2009;301(6):636-650.
- 87. Gunderson EP, Abrams B. Epidemiology of gestational weight gain and body weight changes after pregnancy. *Epidemiol Rev.* 2000;22(2):261-274.
- 88. Rooney BL, Schauberger CW. Excess pregnancy weight gain and long-term obesity: one decade later. *Obstetrics and gynecology.* 2002;100(2):245-252.
- 89. Gilmore LA, Klempel-Donchenko M, Redman LM. Pregnancy as a window to future health: Excessive gestational weight gain and obesity. *Seminars in perinatology*. 2015;39(4):296-303.
- 90. Norman JE, Reynolds RM. The consequences of obesity and excess weight gain in pregnancy. *Proc Nutr Soc.* 2011;70(4):450-456.
- 91. Winkvist A, Brantsaeter AL, Brandhagen M, Haugen M, Meltzer HM, Lissner L. Maternal Prepregnant Body Mass Index and Gestational Weight Gain Are Associated with Initiation and Duration of Breastfeeding among Norwegian Mothers. *J Nutr.* 2015;145(6):1263-1270.

- 92. Verret-Chalifour J, Giguere Y, Forest JC, Croteau J, Zhang P, Marc I. Breastfeeding initiation: impact of obesity in a large Canadian perinatal cohort study. *PloS one*. 2015;10(2):e0117512.
- 93. Thompson LA, Zhang S, Black E, et al. The association of maternal pre-pregnancy body mass index with breastfeeding initiation. *Maternal and child health journal*. 2013;17(10):1842-1851.
- 94. Matthews KA, Croft JB, Liu Y, et al. Health-Related Behaviors by Urban-Rural County Classification United States, 2013. *Morbidity and mortality weekly report Surveillance summaries (Washington, DC: 2002).* 2017;66(5):1-8.
- 95. Hardin-Fanning F, Rayens MK. Food cost disparities in rural communities. *Health promotion practice*. 2015;16(3):383-391.
- 96. Taber DR, Chriqui JF, Quinn CM, Rimkus LM, Chaloupka FJ. Cross-sector analysis of socioeconomic, racial/ethnic, and urban/rural disparities in food policy enactment in the United States. *Health & place*. 2016;42:47-53.
- 97. Lutfiyya MN, Chang LF, Lipsky MS. A cross-sectional study of US rural adults' consumption of fruits and vegetables: do they consume at least five servings daily? *BMC public health*. 2012;12:280.
- 98. Larson NI, Story MT, Nelson MC. Neighborhood environments: disparities in access to healthy foods in the U.S. *American journal of preventive medicine*. 2009;36(1):74-81.
- 99. Bunik M, Clark L, Zimmer LM, et al. Early infant feeding decisions in low-income Latinas. Breastfeeding medicine: the official journal of the Academy of Breastfeeding Medicine. 2006;1(4):225-235.
- 100. Chapman DJ, Perez-Escamilla R. Breastfeeding among minority women: moving from risk factors to interventions. *Advances in nutrition (Bethesda, Md)*. 2012;3(1):95-104.
- 101. Sloand E, Budhathoki C, Junn J, Vo D, Lowe V, Pennington A. Breastfeeding among Latino Families in an Urban Pediatric Office Setting. *Nursing research and practice*. 2016;2016:9278401.
- 102. Mosca L, Mochari-Greenberger H, Dolor RJ, Newby LK, Robb KJ. Twelve-year follow-up of American women's awareness of cardiovascular disease risk and barriers to heart health. *Circ Cardiovasc Qual Outcomes*. 2010;3(2):120-127.
- 103. Bandura A. Human agency in social cognitive theory. *The American psychologist*. 1989;44(9):1175-1184.
- 104. Bandura A. Self-efficacy mechanism in human agency. *The American psychologist*. 1982;37(2):122-147.
- 105. Deci EL, Ryan RM. *The empirical exploration of intrinsic motivational processes*. New York, NY: Academic Press; 1980.
- 106. Deci EL, Ryan RM. A motivational approach to self: Integration in personality. In: Dienstbier R, ed. *Nebraska Symposium on Motivation: Volume 38 Perspectives on Motivation*. Lincoln, NE: University of Nebraska Press; 1991.
- 107. Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. *The American psychologist.* 2000;55(1):68-78.
- 108. Deci EL, Ryan RM. *Intrinsic motivation and self-determination in human behavior*. New York, NY: Plenum; 1985.

- 109. U.S. Department of Health and Human Services and U.S. Department of Agriculture. 2015-2020 Dietary Guidelines for Americans. 8th Edition. December 2015. Available at <a href="http://health.gov/dietaryguidelines/2015/guidelines/">http://health.gov/dietaryguidelines/2015/guidelines/</a>.
- 110. Ingram J, Johnson D, Copeland M, Churchill C, Taylor H. The development of a new breast feeding assessment tool and the relationship with breast feeding self-efficacy. *Midwifery*. 2015;31(1):132-137.
- 111. Horta BL, Victora CG. Long-term effects of breastfeeding. 2013.
- 112. High 5 for Mom & Baby. <a href="http://www.high5kansas.org/">http://www.high5kansas.org/</a>. Accessed April 6, 2016.
- 113. U.S. Department of Health and Human Services' Office on Women's Health. Your Guide to Breastfeeding. Washington DC: Office on Women's Health; 2011:48.
- 114. Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. *Journal of obstetric, gynecologic, and neonatal nursing : JOGNN / NAACOG.* 2003;32(6):734-744.
- 115. Tuthill EL, McGrath JM, Graber M, Cusson RM, Young SL. Breastfeeding Self-efficacy: A Critical Review of Available Instruments. *J Hum Lact.* 2016;32(1):35-45.
- 116. Creedy DK, Dennis CL, Blyth R, Moyle W, Pratt J, De Vries SM. Psychometric characteristics of the breastfeeding self-efficacy scale: data from an Australian sample. *Res Nurs Health*. 2003;26(2):143-152.
- 117. Otsuka K, Taguri M, Dennis CL, et al. Effectiveness of a breastfeeding self-efficacy intervention: do hospital practices make a difference? *Maternal and child health journal*. 2014;18(1):296-306.
- 118. Ainsworth BE, Sternfeld B, Richardson MT, Jackson K. Evaluation of the kaiser physical activity survey in women. *Medicine and science in sports and exercise*. 2000;32(7):1327-1338.
- 119. Schmidt MD, Freedson PS, Pekow P, Roberts D, Sternfeld B, Chasan-Taber L. Validation of the Kaiser Physical Activity Survey in pregnant women. *Medicine and science in sports and exercise*. 2006;38(1):42-50.
- 120. Thompson FE, Subar AF, Smith AF, et al. Fruit and vegetable assessment: performance of 2 new short instruments and a food frequency questionnaire. *J Am Diet Assoc.* 2002;102(12):1764-1772.
- 121. Yaroch AL, Tooze J, Thompson FE, et al. Evaluation of three short dietary instruments to assess fruit and vegetable intake: the National Cancer Institute's food attitudes and behaviors survey. *J Acad Nutr Diet*. 2012;112(10):1570-1577.
- 122. George SM, Thompson FE, Midthune D, et al. Strength of the relationships between three self-reported dietary intake instruments and serum carotenoids: the Observing Energy and Protein Nutrition (OPEN) Study. *Public Health Nutr.* 2012;15(6):1000-1007.
- 123. Dietary Screener Questionnaire in the NHANES 2009-10: Background. <a href="http://epi.grants.cancer.gov/nhanes/dietscreen/">http://epi.grants.cancer.gov/nhanes/dietscreen/</a>. Accessed March 9, 2016.
- 124. Dietary Screener Questionnaire (DSQ) in the NHANES 2009-10: Dietary Factors, Food Items Asked, and Testing Status for DSQ.

  <a href="http://epi.grants.cancer.gov/nhanes/dietscreen/evaluation.html#pub">http://epi.grants.cancer.gov/nhanes/dietscreen/evaluation.html#pub</a>. Accessed March 14, 2016.

- 125. Ruyak SL, Corwin EJ, Lowe NK, Neu M, Boursaw B. Prepregnancy Obesity and a Biobehavioral Predictive Model for Postpartum Depression. *Journal of obstetric, gynecologic, and neonatal nursing : JOGNN / NAACOG.* 2016.
- 126. Records K, Keller C, Coonrod D, et al. Correlates of depressive symptoms after birth for Latinas who are overweight or obese. *Health Care Women Int.* 2015;36(3):356-374.
- 127. Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. *Br J Psychiatry*. 1987;150:782-786.
- 128. Wisner KL, Parry BL, Piontek CM. Clinical practice. Postpartum depression. *N Engl J Med.* 2002;347(3):194-199.
- 129. Gibson J, McKenzie-McHarg K, Shakespeare J, Price J, Gray R. A systematic review of studies validating the Edinburgh Postnatal Depression Scale in antepartum and postpartum women. *Acta Psychiatr Scand.* 2009;119(5):350-364.
- 130. Zou G. A modified poisson regression approach to prospective studies with binary data. *Am J Epidemiol.* 2004;159(7):702-706.